CLINICAL TRIAL: NCT01126671
Title: Clinical Trial of Vitamin D Supplementation in Healthy Adolescents
Brief Title: Vitamin D Supplementation in Healthy Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sarah Pitts, Attending Physician, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-06-0271
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Vitamin D Supplementation
Keywords: vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Vitamin D (Active Comparator): Subjects are randomized to take 200 IU vitamin D3 daily in this arm.
  Interventions: Drug: Supplemental Vitamin D
- High Dose Vitamin D (Active Comparator): Subjects are randomized to take 1000 IU vitamin D3 daily in this arm.
  Interventions: Drug: Supplemental Vitamin D

INTERVENTIONS:
Drug: Supplemental Vitamin D — Subjects were randomized to either take 200 IU of vitamin D or 1000 IU of vitamin D daily for 11 weeks and labs were compared before and after.

SUMMARY:
This double blind, randomized controlled trial compares two supplemental doses of vitamin D in health adolescents.

DETAILED DESCRIPTION:
Vitamin D deficiency is a common problem. Currently, data do not support a recommended vitamin D supplementation dose for health adolescents to maintain normal vitamin D levels. This double blind, randomized controlled 12 week trial compares the use of two supplemental doses of vitamin D in this population.

ELIGIBILITY:
Inclusion Criteria:

* 11-18 years old
* healthy

Exclusion Criteria:

* chronic disease
* use of medication known to effect bone or vitamin D metabolism
* abnormal vitamin D or calcium at screening
* pregnant
* body mass index <5% or >95%

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Putman, MD, Principal Investigator — Childrens Hospital, Boston; Sarah Pitts, MD, Principal Investigator — Childrens Hospital, Boston
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Putman MS, Pitts SA, Milliren CE, Feldman HA, Reinold K, Gordon CM. A randomized clinical trial of vitamin D supplementation in healthy adolescents. J Adolesc Health. 2013 May;52(5):592-8. doi: 10.1016/j.jadohealth.2012.10.270. Epub 2012 Dec 23. PMID 23608721

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Boston Children's Hospital (BCH) Adolescent Medicine Outpatient Program and from the community via flyers, internet postings, and newspaper advertisements. Enrollment began September 1, 2008 and ended March 18, 2011.
Pre-assignment Details: Healthy adolescents, ages 11-19 years, were eligible if clinically healthy, likely to comply with treatment, and not vitamin D deficient.
  Fifty-six patients were enrolled, and two patients were randomized to a treatment group but did not complete a baseline visit and therefore are not included in the analysis.
Groups:
- Low Dose Vitamin D: Subjects in this arm of the study took 200 IU vit D3 daily.
- High Dose Vitamin D: Subjects in this arm of the study took 1000 IU vit D3 daily.
Period: Overall Study
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Started | 26 | 30
Completed | 24 | 29
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 subjects were randomized to a treatment group but did not complete the baseline assessment.
  Participants
    <=18 years | 24 | 26 | 50
    Between 18 and 65 years | 1 | 3 | 4
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.1 (2.2) | 16.1 (2.2) | 16.1 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 4 | 11 | 15
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Baseline 25 Hydroxy Vitamin D (25OHD) Levels
Description: 25OHD will be drawn at baseline prior to starting vitamin D supplementation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 25 | 29
ng/ml | 28.1 (6.2) | 29 (7.3)

2. Primary Outcome: Follow-up 25OHD Levels
Description: After 11weeks of treatment, repeat 25OHD levels will be drawn to assess subject response to vitamin D supplementation.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 25 | 29
ng/ml | 28.9 (7) | 30.1 (6.6)

3. Secondary Outcome: Baseline Assessment of Bone Markers
Description: Bone specific alkaline phosphatase, CTx, and osteocalcin will be assessed at baseline prior to subjects starting vitamin D supplementation
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 25 | 29
ng/ml | 1.4 (0.84) | 1.74 (1.09)

4. Secondary Outcome: Assessment of Bone Markers at Follow-up
Description: After 11 weeks of vitamin D supplementation bone specific alkaline phosphatase, osteocalcin, and CTx will be repeated to see response to therapy.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 25 | 29
ug/L | 31.1 (31.1) | 32.3 (32.3)

ADVERSE EVENTS:
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/29
Other Adverse Events (participants affected / at risk) | 0/25 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes